CLINICAL TRIAL: NCT06965972
Title: Prospective Cohort for the Study of Phenotypic Clusters, Progression Paths and Outcomes of Frailty and Dependence: The Spanish CohorFES
Brief Title: The CohorFES: a Prospective Study of Frailty and Dependence
Acronym: COHORFES
Status: Recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); CIBER on frailty and healthy ageing (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI19/00033
Record Dates: First submitted 2025-04-07; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: Frailty Syndrome
Keywords: COHORFES; Frailty; FTS5
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SERUM, PLASMA, URINE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women and men 65 years old or above visited in the outpatient clinics of participant centers: To stablish the CohorFES, a prospective and observational study based on real population. Patients are recruited from the beginning of the project and followed year on year during all the study time.
  Individuals visited in participant centers and meet inclusion criteria are asked to participate into the study. These individuals are consecutively included to the study after signed the informed consent.

SUMMARY:
Background Frailty has become a major problem for the health system, but also a window of opportunity to fight against disability through preventive strategies focused on the detection and treatment of frailty in all settings. However, no systematic strategies of screening and early detection are available in clinical settings. This project aims to identify clinical and biological phenotypic clusters that drive through the different stages of frailty and to describe the underlying mechanisms of the trajectories leading to disability and the potential for treatment. Moreover, validation of Frailty Trait Scale 5 (FTS5) will be performed as an easy model to be implemented in primary care and hospital scope.

Methods/design A prospective population-based cohort will be stablished for frailty phenotyping (CohorFES). Creation of a CIBERFES Biobank where blood and urine samples from participants of CohortFES are stored for future researches. Demographic and clinical history data, anthropometric measurements, predimed questionnaire, peripheral blood biochemical variables and metabolomics were collected for each participant at baseline and every year until become frailty.

Using cluster partition models (k-means and hierarchical clustering) will group together individuals with similar deficits and characteristics (frailty phenotypes). Then, by using pre-established criteria (gap and silhouette), the proposed clustering solution (belonging to given clusters) will be evaluated. Further, investigators will assess, in a longitudinal fashion, the appearance and accumulation of deficits during the study period and identifying the clusters subgroups with more rapid progression. Results will be applied to establish and compare clusters and trajectories. Finally, frailty phenotypes and patient clusters will be correlated with health outcomes such as the use of health services (both primary and secondary care), hospital admissions, and mortality.

Discussion Information about clinical and biological phenotypic clusters that drive through the different stages of frailty can lead to identify potential targets that could improve the therapeutic management of these patients.

In summary, from a research perspective the project aims to better understanding of the interindividual variability in clinical events that lead to frailty, dependence and finally, to death.

DETAILED DESCRIPTION:
1. Background of the study:

   Frailty is one of the major challenges of the 21st Century, and a top priority for national and international organisms like the WHO (World Health Organization) or the European Parliament. This has put frailty as one of the top priorities in the biomedical research agenda of the European Commission. Frailty is constituted by a physiological state of increased vulnerability and impaired resilience to stressors (i.e. diseases, external agents, drugs tolerability and toxicity) due to the combined effect of the aging process and some chronic diseases which drives to a final stage of dependency and disability with a sharp impact in quality of life, health and social resources consumption, hospitalization and death.

   It is well-known the relevance of frailty, its detection, and management since we are aware about their reversibility, the costs on the health systems, and its potential impact in clinical settings. In a clear contrast with the abundancy of data in non-clinical settings, there is a lack of strong data in the clinical setting where the prevalence of frailty is higher and where the risks for developing its most serious adverse consequences is more likely. There is hence an urgent need for a better screening and diagnosis of frailty, its trajectories and the determinants of these separate trajectories depending upon both the characteristics of frailty in each patient (associated or not with sarcopenia, or cognitive impairment or different clusters of chronic diseases).
2. Review of prior research:

   While the different categories of the syndrome based on the severity of the observed deficits (robust, frail, pre-frail) are quite well defined and characterized from an epidemiological point of view, there is a scarcity of data on the functional pathways between these diagnostic categories (and, among them, disability), and this is especially true in clinical cohorts. This is really shocking considering that one of the most relevant factors, if not the first one, associated with a poor evolution of frailty is to experience an episode of hospitalization.

   The overarching goal of this study is therefore, to identify the critical subgroups of subjects at risk of progression from robustness to prefrailty and frailty and from there to their late stages, and the pathways that mediate this trajectory amongst community-dwelling Spanish subjects.

   Another important issue in this field would be to find an easy tool to identify frailty and factors which could be implemented in our full outpatients list. In addition to the more classical instruments to assess frailty, several groups currently members of CIBER on Frailty and Healthy Ageing (CIBERFES) developed an instrument that overcomes some of the problems raised by the more classical ones. The Frailty Trait Scale-FTS has shown a good predictive capacity for some outcomes in very old patients living in the community. More recently, and as part of an EU-funded project (FRAILTOOLS) we have found that the full version of FTS is able to detect frailty in some clinical settings (Acute Care Geriatric Unit, Geriatric Service outpatient office and Primary Care), with a good predictive capacity for adverse outcomes (death, incident disability, deterioration in SPPB, falls and hospitalization) at 6-12-18 months. However, the full version of FTS, composed of 12 items, takes around 15 minutes, making it unpractical in usual clinical conditions, where the time available by the physician or the nurse is lower. With this fact in mind, a shorter version of only 5 items (the so-called FTS 5) was developed.

   This shorter version takes less time, but more interestingly, FTS 5 offers promising results based upon the sensitivity to detect small changes shown by the full FTS. Finally, the variables that compose the FTS5 (gait velocity, grip strength, BMI, PASE, and balance) can be incorporated into electronic instruments. This has been the case for the electronic frailty index (eFI), developed and validated in the British electronic records based on the Rockwood's frailty model that would allow to assess the frailty profile after to consider 36 items or deficits at the same moment of visit by primary care o hospital physician or the more recent Hospital Frailty Risk Score based on clinical diagnoses that is able to predict death but showing only a fair concordance with the Frailty Phenotype and the Frailty Index.

   The use of easy electronic tools has been useful not only in hospital care but also in routine primary care practice. Moreover, it would be easier to measure the adverse outcomes, including falls, delirium, disability, care home admission, hospitalization and mortality as it has been recently shown.
3. Rationale of study:

Inside this conceptual framework and considering the scarce data available in clinical settings about frailty diagnosis, trajectories and prognosis, the main goal of this project is to stablish a clinical, real-life and prospective cohort (COHORFES) to identify clinical and biological phenotypic clusters that drive through the different stages of frailty and to identify the underlying mechanisms that finally will trigger the disability.

ELIGIBILITY:
Inclusion Criteria:

* women and men 65 years old or above visited in the outpatient clinics of participant centers
* Signed informed consent

Exclusion Criteria:

* Patients in a critical situation of end of live or Barthel scale <60.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants are women and men 65 years old or above visited in the outpatient clinics of participant centers:
  Hospital General Universitario Gregorio Marañón, Madrid Hospital Universitario de Getafe, Madrid Hospital General Universitario de Ciudad Real, Ciudad real Hospital del Mar, Consorci Mar Parc Salut de Barcelona, Barcelona Complejo Hospitalario Universitario de Albacete, Albacete Fundación del Hospital Nacional de Parapléjicos, Toledo
  These participants are included in the COHORFES
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Fried phenotype | Through study completion, an average of 5 years
  Frailty measure
Frailty Trait Scale 5 ítems: 1.- walking speed test, 2.- grip strength, 3.- Physical Activity, 4- Body Mass Index (BMI), 5.- progressive Romberg test. Point 1 to 5 are combined to report the frailty trait scale | Through study completion, an average of 5 years
  Frailty measure
Electronic Frailty index | Through study completion, an average of 5 years
  Frailty measure

SECONDARY OUTCOMES:
Bone Mineral Density | Through study completion, an average of 5 years
  Bone Mineral Density measured using a Dual-Energy X-Ray Analysis (DXA) device (Hologic Horizon Wi, Hologic®).
Abnormal peripheral blood biochemistry | Through study completion, an average of 5 years
  Detection of anormal values of the following parameters (y/n):
  * Leukocytes ml/mmc
  * Red blood cells ml/mmc
  * Hemoglobin g/dl
  * Hematocrit %
  * Red blood cell distribution width %
  * Platelets ml/mmc
  * Vitamin D ng/ml
  * TSH nmol/l
  * Glucose mg/dl
  * Glycated hemoglobin (diabetics only) %
  * Creatinine mg/dl
  * Sodium meq/dl
  * Potassium meq/dl
  * Calcium mg/dl
  * Phosphorus mg/dl
  * GPT u/l
  * GOT u/l
  * Phosphatase alkaline u/l
  * Total proteins g/dl
  * Albumin g/dl
  * Prealbumin mg/dl
  * Cholesterol mg/dl
  * Triglycerides mg/dl
  * HDL mg/dl
  * LDL mg/dl
  * C-reactive protein mg/ml
  These parameters are combined with the final outcome: abnormal biochemistry (y/n)
Age | baseline
  Age in years
Date of Birth | baseline
  Date (dd/mm/yyyy)
Sex | baseline
  sex (Male or Female)
Living situation | baseline
  Living situation: Alone or accompanied
Educational level | baseline
  Educational level: number of years in the school and college
All-cause mortality. | From baseline until the date of death from any cause, an average of 5 years
  mortality during study follow-up (y/n)
Condition diagnosis | Through study completion, an average of 5 years
  New condition diagnosis during follow-up (for ex. diagnosis of cancer, fracture, dementia, etc)
Usual treatments | Through study completion, an average of 5 years
  treatments being taken by the patient
Pharmacy use | Through study completion, an average of 5 years
  number of different drugs being taken by the patient
Loss of weight | Through study completion, an average of 5 years
  Loss of weight in the last year in grams
Geriatric Depression Scale | Through study completion, an average of 5 years
  Geriatric Depression Scale: 15 items (y/n) were combined to report GDS
Barthel Index | Through study completion, an average of 5 years
  Barthel Index: measure of functional disability
Lawton-Brody Instrumental Activities of Daily Living Scale | Through study completion, an average of 5 years
  to assess independent living skills. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning).
Pfeiffer test | Through study completion, an average of 5 years
  test of 10 questions used to assess a person's cognitive status
Predimed questionnaire | Through study completion, an average of 5 years
  The adherence of participants to the Mediterranean diet will be assessed through the 14-item Mediterranean diet adherence screener (MEDAS) validated for the Spanish population in a phone interview with the participant
Healthcare resource use | Through study completion, an average of 5 years
  number of medical care consultations
Non-elective hospital admissions | Through study completion, an average of 5 years
  Number of admissions in a Hospital

OTHER OUTCOMES:
Metabolomics | Through study completion, an average of 5 years
  Quantitative metabolomics approach applied to analyze plasma samples using liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS). It is defined as altered metaboloma (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Nogues, PhD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar Research Institute, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Once the project is completed and after the necessary embargo periods, de-identified data will be shared with the research community upon request to the PI of the study. Intellectual property rights or sensitive data will be handled in accordance with the EU General Data Protection Regulation (GDPR). As this is a prospective observational cohort with long-term clinical data collection, the data will be deposited in the IMIM repository and shared upon request to the research group responsible for the data.
  Data dissemination will take place through academic journals and conference presentations.
Time Frame: from 1/1/2035 to 31/12/2050
Access Criteria: All researcher can request to the Hospital del Mar Research Institute the anomyzed IPD from 1/1/2035

REFERENCES:
- [Result] Stow D, Matthews FE, Barclay S, Iliffe S, Clegg A, De Biase S, Robinson L, Hanratty B. Evaluating frailty scores to predict mortality in older adults using data from population based electronic health records: case control study. Age Ageing. 2018 Jul 1;47(4):564-569. doi: 10.1093/ageing/afy022. PMID 29546362
- [Result] Gilbert T, Neuburger J, Kraindler J, Keeble E, Smith P, Ariti C, Arora S, Street A, Parker S, Roberts HC, Bardsley M, Conroy S. Development and validation of a Hospital Frailty Risk Score focusing on older people in acute care settings using electronic hospital records: an observational study. Lancet. 2018 May 5;391(10132):1775-1782. doi: 10.1016/S0140-6736(18)30668-8. Epub 2018 Apr 26. PMID 29706364
- [Result] Clegg A, Bates C, Young J, Ryan R, Nichols L, Teale EA, Mohammed MA, Parry J, Marshall T. Development and validation of an electronic frailty index using routine primary care electronic health record data. Age Ageing. 2018 Mar 1;47(2):319. doi: 10.1093/ageing/afx001. No abstract available. PMID 28100452
- [Result] Garcia-Garcia FJ, Carnicero JA, Losa-Reyna J, Alfaro-Acha A, Castillo-Gallego C, Rosado-Artalejo C, Gutierrrez-Avila G, Rodriguez-Manas L. Frailty Trait Scale-Short Form: A Frailty Instrument for Clinical Practice. J Am Med Dir Assoc. 2020 Sep;21(9):1260-1266.e2. doi: 10.1016/j.jamda.2019.12.008. Epub 2020 Jan 29. PMID 32005416
- [Result] Checa-Lopez M, Oviedo-Briones M, Pardo-Gomez A, Gonzales-Turin J, Guevara-Guevara T, Carnicero JA, Alamo-Ascencio S, Landi F, Cesari M, Grodzicki T, Rodriguez-Manas L; FRAILTOOLS consortium. FRAILTOOLS study protocol: a comprehensive validation of frailty assessment tools to screen and diagnose frailty in different clinical and social settings and to provide instruments for integrated care in older adults. BMC Geriatr. 2019 Mar 18;19(1):86. doi: 10.1186/s12877-019-1042-1. PMID 30885132
- [Result] Garcia-Garcia FJ, Carcaillon L, Fernandez-Tresguerres J, Alfaro A, Larrion JL, Castillo C, Rodriguez-Manas L. A new operational definition of frailty: the Frailty Trait Scale. J Am Med Dir Assoc. 2014 May;15(5):371.e7-371.e13. doi: 10.1016/j.jamda.2014.01.004. Epub 2014 Mar 2. PMID 24598478
- [Result] Gill TM, Gahbauer EA, Han L, Allore HG. The relationship between intervening hospitalizations and transitions between frailty states. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1238-43. doi: 10.1093/gerona/glr142. Epub 2011 Aug 17. PMID 21852286
- [Result] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Rodriguez-Manas L, Rodriguez-Artalejo F, Sinclair AJ. The Third Transition: The Clinical Evolution Oriented to the Contemporary Older Patient. J Am Med Dir Assoc. 2017 Jan;18(1):8-9. doi: 10.1016/j.jamda.2016.10.005. Epub 2016 Nov 22. No abstract available. PMID 27887892
- [Result] Rodriguez-Manas L, Fried LP. Frailty in the clinical scenario. Lancet. 2015 Feb 14;385(9968):e7-e9. doi: 10.1016/S0140-6736(14)61595-6. Epub 2014 Nov 6. No abstract available. PMID 25468154
- [Result] Sirven N, Rapp T. The cost of frailty in France. Eur J Health Econ. 2017 Mar;18(2):243-253. doi: 10.1007/s10198-016-0772-7. Epub 2016 Feb 25. PMID 26914932
- [Result] Trombetti A, Hars M, Hsu FC, Reid KF, Church TS, Gill TM, King AC, Liu CK, Manini TM, McDermott MM, Newman AB, Rejeski WJ, Guralnik JM, Pahor M, Fielding RA; LIFE Study Investigators. Effect of Physical Activity on Frailty: Secondary Analysis of a Randomized Controlled Trial. Ann Intern Med. 2018 Mar 6;168(5):309-316. doi: 10.7326/M16-2011. Epub 2018 Jan 9. PMID 29310138
- [Result] Rodriguez-Manas L, Feart C, Mann G, Vina J, Chatterji S, Chodzko-Zajko W, Gonzalez-Colaco Harmand M, Bergman H, Carcaillon L, Nicholson C, Scuteri A, Sinclair A, Pelaez M, Van der Cammen T, Beland F, Bickenbach J, Delamarche P, Ferrucci L, Fried LP, Gutierrez-Robledo LM, Rockwood K, Rodriguez Artalejo F, Serviddio G, Vega E; FOD-CC group (Appendix 1). Searching for an operational definition of frailty: a Delphi method based consensus statement: the frailty operative definition-consensus conference project. J Gerontol A Biol Sci Med Sci. 2013 Jan;68(1):62-7. doi: 10.1093/gerona/gls119. Epub 2012 Apr 16. PMID 22511289
- [Result] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209